CLINICAL TRIAL: NCT07252895
Title: Walking Ability of Patients With Multiple Sclerosis Using the EXOPULSE Suit: Randomized Controlled Crossover Trial
Brief Title: EXOPULSE Suit and Walking Ability of Patients With Multiple Sclerosis
Acronym: EXO-MOBILITY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Otto Bock France SNC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: BP-11-PT-010
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; neuromodulation; suit; walking ability; multi-site electrical stimulation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Each participant is his/her own control
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXOPULSE Suit Active then EXOPUSLE Suit sham (Other): The participant is fist using the EXOPULSE Suit in Active mode for 4 weeks, then he has a 4-weeks wash-out period, then he is using the EXOPULSE Suit in a sham mode for 4 weeks.
  Interventions: Device: EXOPULSE Suit in Active mode; Device: EXOPULSE Suit in Sham mode
- EXOPULSE Suit in sham mode then EXOPULSE Suit in Active mode (Other): The participant is first using the EXOPUISE Suit in sham mode for 4 weeks, then he has a 4-weeks wash-out phase, the he is using the EXOPULSE Suit in Active mode for 4 weeks.
  Interventions: Device: EXOPULSE Suit in Active mode; Device: EXOPULSE Suit in Sham mode

INTERVENTIONS:
Device: EXOPULSE Suit in Active mode — The EXOPULSE Suit in Active mode stimulates the targeted muscles during the whole 60-minutes cession
Device: EXOPULSE Suit in Sham mode — The EXOPULSE Suit in Sham mode stimulates the targeted muscles during the first minute of the cession then is off during the 59 minutes left.

SUMMARY:
The EXOPULSE Suit is medical device composed of 50 electrods that can stimulate up to 43 main muscle groups of the body. The multisite electrical stimulation relaxes tens and spastic muscles, thus enhance mobility and balance. This non-invasive body garment is a home-use device which should be used for 1 hour every other day.

This research aims at confirming the benefits of EXOPULSE Suit in persons with Multiple Sclerosis, including the walking ability.

DETAILED DESCRIPTION:
Lower limb function is perceived as being essential by persons with multiple sclerosis (pwMS). The loss of walking ability is a major physical manifestation among MS patients with EDSS between 4 and 7, that negatively impacts activities of daily living and employment. Different therapeutic means can be proposed to maintain or improve mobility such as rehabilitation, that is an essential and irreplaceable element of the patient's journey, or the im-plementation of treatments aiming at decreasing symptoms like spasticity, fatigue or pain.

The only treatment exclusively aiming at improving walking ability is the Fampridine medicine . Nevertheless, all patients cannot benefit from it due to contra-indications, side effects or because they are not responders or no longer responders to Fampridine. Some others simply do not want to take drugs.

The EXOPULSE Suit is a class IIa certified electrical medical device composed of 50 electrods that can stimulate up to 43 main muscle groups of the body. The multi-site electrical stimulation relaxes tens and spastic muscles, thus enhance mobility and balance. This non-invasive body garment is a home-use device which should be used for 1 hour every other day.

EXOPULSE Suit could be an alternative for improving walking ability of patients who cannot be treated with Fampridine medicine.

This research aims at confirming the benefits of EXOPULSE Suit in pwMS. It should highlight an improved walking ability with the EXOPULSE Suit when compared to sham condition.

ELIGIBILITY:
Inclusion Criteria:

* Person with a clear Multiple Sclerosis diagnosis according to the 2017 revision of the McDonald criteria since at least 3 months.
* Person with an Expanded Disability Status Scale (EDSS) score ≥ 4 and ≤ 6
* Person with stable walking ability for at least two weeks prior to the inclusion visit (variation at the MSWS-12 questionnaire < 8/100 points)
* Person not treated with fampridine due to contra-indication or adverse events or not respondent or no longer respondent or reluctant to taking drugs
* Person with spasticity at the lower limb(s), attested by a Modified Ashworth Scale ≥ 1+ of at least one of the following muscle groups: quadriceps, hamstrings, triceps surae, tibialis anterior
* Person who never tried EXOPULSE SUIT

Exclusion Criteria:

* Person under 18 years old
* Person having a contraindication to using EXOPULSE SUIT
* Person using an electronic life-support equipment, e.g. pacemakers or hight-frequency surgical equipment and person using an ECG equipment
* Person affected by other somatic or neuropsychiatric diagnoses (e.g., arrhythmias, uncontrolled epilepsy, diseases causing osteoarticular and muscular pain).
* Person with relapses over the last 3 months before the inclusion
* Person who had a modification of his/her medical treatments of the multiple sclerosis or related to motor performance over the last 3 months before the inclusion
* Person who had a new medical treatment of the multiple sclerosis or related to motor performance over the last 3 months before the inclusion
* Person who had an injection of botulinum toxin in at least one of the main muscle groups of the lower limbs over the last 4 months before the inclusion
* Person planning to use a new medical device during the study (ex: ankle-foot orthosis…)
* Person undergoing or planning to undergo an intensive rehabilitation phase
* Person that is part of another study
* Person who cannot be fitted with EXOPULSE SUIT due to inexistent Suitable size of the Suit (eg: BMI>35; user height < 100 cm or > 205cm)
* Person who does not have a smartphone or who cannot or does not want to use his/her smartphone for operating the EXOPULSE App
* Person not available to undergo all medical visits during the study
* Person unable to understand verbal and written instructions in french
* Pregnant person
* Persons under juridical protection
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
The Multiple Sclerosis Walking Scale 12 (MSWS-12) | 28 days
  The Multiple Sclerosis Walking Scale 12 (MSWS-12) is a 12-item assessment tool designed to measure the impact of multiple sclerosis (MS) symptoms on patients' walking and balance ability, through a series of questions about various daily activities performed over the previous two weeks. Patients are asked to rate the impact of MS on their mobility using a five-point Likert scale, ranging from 1, indicating "no im-pact", to 5, meaning "extremely significant impact". The final score is obtained by adding the responses to the 12 questions (with a sum ranging from 12 to 60). This sum is then converted to a scale of 0 to 100, where a higher score reflects a greater impact of symptoms on the patient's walking ability.

SECONDARY OUTCOMES:
10 Meters Walk Test (10MWT) | 28 days
  The 10MWT is a performance measure that assesses walking speed in meters per second over a short dis-tance. A high score indicates a fast-walking speed. At a comfortable speed, the patient is asked to walk over 10 meters, plus 2 meters at the beginning and at the end for acceleration and deceleration.
2-minute Walk Test (2MWT) | 28 days
  The 2-minute Walk test is a measurement of endurance that assesses the maximum walking distance over 2 minutes. A long walking distance reflects good endurance.
Timed-up and go Test (TUG) | 28 days
  The Timed Up and Go (TUG) test is a validated tool in people with MS to assess functional mobility. It measures the time it takes a person to get up from a chair (without the help of the hands), walk 3 meters, turn around a cone / mark on the floor, return to the chair, and sit back down. Patients are instructed to complete the course as safely and quickly as possible. If needed, patients are allowed to use assistive devices while performing the task. They are given 2 trials to complete the TUG test and the computed time across the 2 trials is the final score.
  A high value reflects an increased risk of falling.
Visual Analog Scale - Fatigue (VAS - Fatigue) | 28 days
  The VAS is a measurement tool where the patient rates his fatigue level by marking a point on a 10 cm line that represents a continuum between "no fatigue" and "worst possible fatigue". The measurement (in mm) between the left end of the line and the mark done by the patient represents the level of fatigue perceived by the patient. The score is then expressed by a note between 0 and 10, 10 being the worst pos-sible fatigue.
The Modified Ashworth Scale (MAS) | 28 days
  The Modified Ashworth Scale (MAS) is a revised version of the original Ash-worth Scale that measures spasticity in patients with lesions to the central nervous system.
  MAS measures the increase in muscle tone by assigning a grade of spasticity from 0 to 4. The grade is assigned by moving a joint/muscle through a high velocity quick stretch.
  MAS grades:
  0 : No increase in muscle tone
  1 : Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  1+ : Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM (range of movement) 2 : More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved 3 : Considerable increase in muscle tone passive, movement difficult 4 : Affected part(s) rigid in flexion or extension
The Multiple Sclerosis Impact Scale 29-items (MSIS-29) | 28 days
  The Multiple Sclerosis Impact Scale 29-items (MSIS-29) is 29-items' self-questionnaires that measure the physical and psychological impact of MS on day-to-day life in the past two weeks. . It comprises 20 items associated with a physical scale and a 9-items scale with a psychological scale. Each item has 5 response options going from 1 "not at all" to 5 "extremely". Each of the two scales are scored by summing the response across items, then converting to a 0-100 scale where 100 indicates a greater impact of disease on daily function.
  The physical impact score is computed by summing items number 1-20 inclusive. This score can then be transformed to a score on a scale of 0 -100 using this formula: (100*(observed score-20))/(100-20).
  The psychological impact score is computed by summing items number 21-29 inclusive. This score can then be transformed to a score on a scale of 0 -100 using this formula: (100*(observed score-9)/(45-9).
The EuroQol - 5 Dimensions -5 levels (EQ-5D-5L) | 28 days
  The EuroQol - 5 Dimensions -5 levels (EQ-5D-5L) is a scale developed by the EuroQol group that assesses quality of life through 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxie-ty/depression. Each dimension has 5 levels going from "no problems" to "extreme problems". Health status can be defined by an index value that goes between 0 and 1. It expresses how is the health status, according to preferences of the general population of a given country. Health status is also expressed by the EQ VAS (Visual Analogue Scale). The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labeled 'The best health you can imagine' and 'The worst health you can imagine'. VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgment.
Visual Analog Scale - Pain (VAS - Pain) | 28 days
  The VAS is a measurement tool where the patient rates his perceived general pain level by marking a point on a 10 cm line that represents a continuum between "no pain" and "worst possible pain". The measurement (in mm) between the left end of the line and the mark done by the patient represents the level of pain perceived by the patient. The score is then expressed by a note between 0 and 10, 10 being the worst possible pain.

OTHER OUTCOMES:
Feeling during the stimulation | 28 days
  4 additional questions related to the feeling during the stimulation will be asked: pain, tingling, burning, fatigue.
  Data considered are with EXOPULSE Suit in active mode.
Satisfaction with the suit | 28 days
  4 additional questions related to the satisfaction with the suit will be asked: ease for putting on and off, ease of use, comfort with the suit, efficacy.
  Data considered are with EXOPULSE Suit in active mode.

CONTACTS AND LOCATIONS:
Overall Officials: Samar AYACHE, Pr, Study Chair — CHU Henri Mondor; Djamel BENSMAIL, Pr, Study Chair — Hôpital Raymond Poincaré; Jérôme DE SEZE, Pr, Study Chair — Hôpital de Hautepierre; Volker LIMMROTH, Pr, Study Chair — Klinik für Neurologie Köln-Merheim
Locations (11):
- France (11):
  - Centre Jacques Calvé Fondation Hopale, Berck
  - CHU Henri Mondor, Créteil
  - CHU Dijon, Dijon
  - Clinique Verdaich, Gaillac-Toulza
  - Hôpital Raymond-Poincaré, Garches
  - Hopital Saint Philibert, Lomme
  - Centre Médical Germaine REVEL, Lyon
  - Hôpital L'Archet, Nice
  - Pole MPR Saint Hélier, Rennes
  - Hôpital Henry Gabrielle, Saint-Genis-Laval
  - Hôpital de Hautepierre, Strasbourg

IPD SHARING:
Plan to Share IPD: No